CLINICAL TRIAL: NCT05221736
Title: Comparison Between Ultrasound-Guided Ethanol Sclerotherapy (UGES) & Surgical Excision in Management of Warthin Tumor of Parotid Gland.
Brief Title: Management of Warthin Tumor of Parotid Gland.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, kerolos nashaat hosny, assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Warthin tumor of parotid gland
Record Dates: First submitted 2022-01-07; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Warthin's Tumor of Parotid Gland

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Warthin tumor in parotid tumor (Experimental): Comparison between Ultrasound-Guided Ethanol Sclerotherapy (UGES) & surgical excision in management of warthin tumor of parotid gland.
  Interventions: Procedure: Ultrasound-Guided Ethanol Sclerotherapy (UGES)

INTERVENTIONS:
Procedure: Ultrasound-Guided Ethanol Sclerotherapy (UGES) — Comparison between Ultrasound-Guided Ethanol Sclerotherapy (UGES) & surgical excision in management of warthin tumor of parotid gland.
  Other Names: Surgical excision

SUMMARY:
Comparison between Ultrasound-Guided Ethanol Sclerotherapy (UGES) & surgical excision in management of warthin tumor of parotid gland.

DETAILED DESCRIPTION:
Warthin tumor (also known as cystadenolymphoma), is a benign and frequent salivary gland neoplasm.

It represents about 2% to 15% of all primary epithelial tumors of the parotid gland.

Warthin tumor is histologically characterized by a dense lymphoid stroma and a double layer of oncocytic epithelium with a papillary and cystic architectural pattern.

Its etiology: remains controversial. Incidence: It is the second most frequent benign neoplasm of the salivary glands after pleomorphic adenoma. Pathophysiology: Initially, Hildebrand proposed that the lesion may be remnants of the branchial pouches and a variant of the lateral cervical cyst. Later, Albrech and Artz proposed the heterotropic origin of Warthin tumor from the neoplastic proliferation of salivary gland ducts present within intra- or para-parotid nodes. Histopathology: Grossly, Warthin tumor is a well-circumscribed spherical to oval mass. On cut section, there are solid areas and multiple cysts with papillary projections.

Cytology: Smears characteristically show oncocytic epithelial cells without atypia admixed with polymorphous lymphocytes and cellular debris.

Microscopic Findings: Warthin tumors are composed of varying proportions of papillary- cystic structures lined by oncocytic epithelial cells and a lymphoid stroma with germinal centers.

Clinically, Warthin tumor presents as a rounded or an ovoid nodular painless, slow-growing, fluctuant to firm at palpation. It can be unilateral, bilateral, or multicentric and is asymptomatic in 90% of cases.

Prognosis: Warthin's tumor has a favorable prognosis and almost never recurs. Malignant degeneration of Warthin tumor is very rare.

Complications:

Local Recurrence; The local recurrence rate is low; when recurrence does occur, it is probably due to multifocal tumors or inadequate excision.

Malignant Transformation; Malignant transformation in a Warthin tumor is extremely rare. The most frequent histological types of malignant transformation in a Warthin tumor are mucoepidermoid carcinoma, squamous cell carcinoma, undifferentiated carcinoma, oncocytic adenocarcinoma, and adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* All new cases presented with benign parotid cyst and diagnosed as Warthin tumour in the parotid gland.

Exclusion Criteria:

* Other Parotid gland tumours e.g. solid tumours, malignant tumours and other suspicious tumours.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Primary (main): | 1 year
  Rate of curability in each group

SECONDARY OUTCOMES:
Secondary (subsidiary): | 1 week
  Rate of facial nerve injury in each group

CONTACTS AND LOCATIONS:
Overall Officials: Hamdan S. Abbas, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
age, sex , clinical diagnosis
Supporting Information: Study Protocol, SAP
Time Frame: 3 years
Access Criteria: age, sex , clinical diagnosis